CLINICAL TRIAL: NCT06293092
Title: Intradialytic Aerobic Versus Resistive Exercises on Immunity Response in Patients With Chronic Kidney Disease
Brief Title: Effect of Intradialytic Exercises in Chronic Kidney Disease Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Hazem Mohamed Yasin Abbas, physiotherapist, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P.T.REC/012/004008
Record Dates: First submitted 2024-02-13; First posted 2024-03-05 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-03

CONDITIONS: Chronic Kidney Disease stage3
Keywords: Exercise; Dialysis; Kidney Failure; Chronic
MeSH Terms: conditions — Motor Activity; Renal Insufficiency; Bronchiolitis Obliterans Syndrome

STUDY DESIGN:
Intervention Model Description: control group receive medical treatment only ,first study group receive medical treatment and intradialytic aerobic exercise , second study group receive medical treatment and intradialytic resistive exercise
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- control group C (Experimental): receive hemodialysis sessions
  Interventions: Device: hemodialysis sessions
- study group A aerobic exercise (Experimental): receive hemodialysis sessions and intradialytic aerobic exercise
  Interventions: Device: leg pedaling cycling device; Device: hemodialysis sessions
- study group B resistive exercise (Experimental): receive hemodialysis sessions and intradialytic resistive exercise
  Interventions: Device: sand bags; Device: hemodialysis sessions

INTERVENTIONS:
Device: leg pedaling cycling device — Intradialytic aerobic cycling exercise program ,each patient will receive the treatment program three times per week for three months.
  Arms: study group A aerobic exercise
Device: sand bags — Intradialytic resistive exercise program , each patient will receive the treatment program three times per week for three months.
  Arms: study group B resistive exercise
Device: hemodialysis sessions — hemodialysis sessions ,each patient will receive the treatment program three times per week for three months.

SUMMARY:
the purpose of this study is to compare between intradialytic aerobic versus resistive exercises on immunity response in patients with chronic kidney disease.

DETAILED DESCRIPTION:
The patients of this study will randomly assigned into three equal groups (n=20)

1. Study Group A (20 patients) will receive intradialytic aerobic exercise and medical treatment.
2. Study Group B (20 patients) will receive intradialytic resistive exercise and medical treatment.
3. Control Group C (20 patients) will receive medical treatment only (HD session and drugs) Each patient will receive the treatment program three times per week for three months.

ELIGIBILITY:
Inclusion Criteria:

* Sixty men chronic kidney disease (grade III RF). They received regular hemodialysis sessions at least one year ago, each one for four hours, three times per week.
* They had a history of type II Diabetes more than five years.
* Their age will be ranged from 50-60 years old.
* They are Fit for exercise by functional assessment using six minute walk test.
* Their Hemoglobin level more than 10 g\dl.
* Their Body Mass Index (BMI) will be ranged from "18.5" to "24.9".

Exclusion Criteria:

* Severe cardiac disorders.
* Severe orthopedic problems (for example fractures).
* Hepatic encephalopathy.
* Preexisting neuromuscular diseases (e.g. myasthenia gravis). •Severe chest diseases.
* Spinal cord injuries involved the phrenic nerve.
* Uncontrolled diabetes or hypertension
* Patients receiving inefficient hemodialysis session.
* Patients with other cause for inflammation e.g. malignancy and autoimmune disease.
* Active bleeding as alveolar hemorrhage, hemoptysis.
* Physical limitation that would limit cycling.

Ages: 50 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2022-04-30 (Actual); Primary Completion 2023-10-30 (Actual); Study Completion 2024-01-30 (Actual)

PRIMARY OUTCOMES:
Concentration of immunoglobulin g | baseline , 12 weeks for each patient
  measured by mg/dl
Total leukocyte count | baseline , 12 weeks for each patient
  measured by (cell/mcl)****1000
lymphocyte count | baseline , 12 weeks for each patient
  measured by (cell/mcl)****1000
neutrophil count | baseline , 12 weeks for each patient
  measured by (cell/mcl)****1000
Concentration of HbA1c | baseline , 12 weeks for each patient
  measured by percentage of blood sugar last 3 months

SECONDARY OUTCOMES:
hemoglobin concentration | baseline , 12 weeks for each patient
  measured by (g/dl)
thrombocytes count | baseline , 12 weeks for each patient
  measured by (cell/mcl)****1000
diastolic blood pressure | baseline , 12 weeks for each patient
  measured by mmHg
Systolic blood pressure | baseline , 12 weeks for each patient
  measured by mmHg
six minute walk test | baseline , 12 weeks for each patient
  measured by meter
(KDQOL-SFTM) questionnaire | baseline , 12 weeks for each patient
  measured by scoring a score-value from 0 (worst health status) to 100 (best health status) was obtained

CONTACTS AND LOCATIONS:
Locations (1):
- Fayoum hospital, Al Fayyum, Egypt